CLINICAL TRIAL: NCT02751918
Title: An Open-label Phase Ib Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Maximum Tolerated Dose of Anetumab Ravtansine in Combination With Pegylated Liposomal Doxorubicin 30 mg/m2 Given Every 3 Weeks in Subjects With Mesothelin-expressing Platinum-resistant Recurrent Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Phase Ib Study of Anetumab Ravtansine in Combination With Pegylated Liposomal Doxorubicin in Patients With Recurrent Mesothelin-expressing Platinum-resistant Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18326
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Ovarian Neoplasms
Keywords: Mesothelin-expressing platinum-resistant cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — anetumab ravtansine; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Anetumab ravtansine (Experimental): Anetumab ravtansine in combination with pegylated liposomal doxorubicin in subjects with mesothelin-expressing platinum-resistant recurrent ovarian, fallopian tube, or primary peritoneal cancer. Increase/Decrease of Anetumab ravtansine until maximum tolerated dose identified.
  Interventions: Drug: Anetumab ravtansine (BAY94-9343); Drug: Pegylated Liposomal Doxorubicin

INTERVENTIONS:
Drug: Anetumab ravtansine (BAY94-9343) — Anetumab ravtansine will be administered on Day 1 of every 21-day treatment cycle.
Drug: Pegylated Liposomal Doxorubicin — Pegylated liposomal doxoribicin will be administered on Day 1 of every 21-day treatment cycle.

SUMMARY:
Anetumab ravtansine is developed for the treatment of patients with recurrent platinum-resistant ovarian cancer. The purpose of the proposed trial is to identify the maximum tolerated dose of anetumab ravtansine that could be safely combined with pegylated liposomal doxorubicin in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with locally invasive or metastatic, epithelial ovarian, fallopian tube, or primary peritoneal cancer
* Subjects must provide samples of tumor tissue
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Subjects with low-grade ovarian, fallopian tube, or Primary peritoneal cancer
* Women who are pregnant or breast feeding
* Subjects who have an active hepatitis B virus or hepatitis C virus infection requiring treatment as defined in the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of Anetumab ravtansine in combination with pegylated liposomal doxorubicin when given every three weeks | Up to 6 months, minimum: 1 cycle (=21days)
  MTD is defined as the highest dose of anetumab ravtansine administered in combination with pegylated liposomal doxorubicin that can be given such that not more than 1 of 6 subjects at a given dose level experiences a dose-limiting toxicity (DLT).
Incidence of serious and non-serious adverse events (AEs) | Up to 6 months

SECONDARY OUTCOMES:
AUC (area under the plasma concentration vs. time curve from zero to infinity after single (first) dose) of Anetumab ravtansine analytes (Antibody drug conjugates, Total Antibody, metabolites DM4, and DM4-Me) | At pre-dose, 0.5h, 1h, 1.5h, 2h, 3h, 5h, 8h, 24h, 48h, 168h, 336h and 504h post-dose, beginning on day 1 of cycle 1
AUC(0-tlast) (AUC from time zero to the last data point > lower limit of quantification) of Anetumab ravtansine analytes (Antibody drug conjugates, Total Antibody, metabolites DM4, and DM4-Me) | At pre-dose, 0.5h, 1h, 1.5h, 2h, 3h, 5h, 8h, 24h, 48h, 168h, 336h and 504h post-dose, beginning on day 1 of cycle 1
Cmax (maximum drug concentration in plasma after first dose administration) of Anetumab ravtansine analytes (Antibody drug conjugates, Total Antibody, metabolites DM4, and DM4-Me) | At pre-dose, 0.5h, 1h, 1.5h, 2h, 3h, 5h, 8h, 24h, 48h, 168h, 336h and 504h post-dose, beginning on day 1 of cycle 1
AUC of total pegylated liposomal doxorubicin | At pre-dose, 0.5h, 1h, 2h, 3h, 6h, 8h, 22h, 46h, and 166h post-dose , beginning on day 1 of cycle 1
AUC(0-tlast) of total pegylated liposomal doxorubicin | At pre-dose, 0.5h, 1h, 2h, 3h, 6h, 8h, 22h, 46h, and 166h post-dose , beginning on day 1 of cycle 1
Cmax of total pegylated liposomal doxorubicin | At pre-dose, 0.5h, 1h, 2h, 3h, 6h, 8h, 22h, 46h, and 166h post-dose, beginning on day 1 of cycle 1
Incidence of patients with CR, PR, SD or PD according to RECIST 1.1 | Up to 17 months or until discontinuation of study, whichever comes first
  CR (complete response) PR (partial response) SD (stable disease) PD (progressive disease)
Incidence of positive anti-drug antibody titer | Up to 17 months or until discontinuation of study, whichever comes first
Incidence of positive neutralizing antibody titer | Up to 17 months or until discontinuation of study, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- United States (3):
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
- UZ Leuven Gasthuisberg, Leuven, Belgium
- The Institute of Oncology, Chisinau, Moldova
- Spain (4):
  - Ciutat Sanitària i Universitaria de la Vall d'Hebron, Barcelona
  - Clinica Universidad de Navarra CUN en Madrid, Madrid
  - Clínica Universidad de Navarra CUN, Pamplona
  - Instituto Valenciano de Oncología, Valencia

REFERENCES:
- [Derived] Santin AD, Vergote I, Gonzalez-Martin A, Moore K, Oaknin A, Romero I, Diab S, Copeland LJ, Monk BJ, Coleman RL, Herzog TJ, Siegel J, Kasten L, Schlicker A, Schulz A, Kochert K, Walter AO, Childs BH, Elbi C, Bulat I. Safety and activity of anti-mesothelin antibody-drug conjugate anetumab ravtansine in combination with pegylated-liposomal doxorubicin in platinum-resistant ovarian cancer: multicenter, phase Ib dose escalation and expansion study. Int J Gynecol Cancer. 2023 Apr 3;33(4):562-570. doi: 10.1136/ijgc-2022-003927. PMID 36564099